CLINICAL TRIAL: NCT01611181
Title: Iron Substitution After Total Knee Arthroplasty - a Randomized Study
Brief Title: Iron Substitution After Total Knee Arthroplasty
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VN 2004/30
Record Dates: First submitted 2012-05-29; First posted 2012-06-04 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Haemodynamic Rebound
Keywords: Iron supplementation; Iron deficiency; Hip arthroplasty; Knee arthroplasty
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hemoboost (iron supplementation) (Active Comparator): A registered natural product containing specially haemolysed haemoglobin and iron dextran.
  Interventions: Drug: Hemoboost
- Kräuterblut (iron supplementation) (Active Comparator): A registered natural product made from a number of herbs with ferrous gluconate as the active substance.
  Interventions: Drug: Kräuterblut
- Ferrofumerat (iron supplementation) (Active Comparator): Ferrous sulphate
  Interventions: Drug: Ferrofumerat

INTERVENTIONS:
Drug: Hemoboost — 200 mg specially processed haemoglobin and 30 mg iron dextran equivalent to 10.5 mg organically bound iron in 1 tablet twice daily.
  Other Names: No other names.
  Arms: Hemoboost (iron supplementation)
Drug: Kräuterblut — 40 mg iron, 20 ml twice daily.
  Other Names: No other names.
  Arms: Kräuterblut (iron supplementation)
Drug: Ferrofumerat — 200 mg ferrous sulphate as 1 tablet twice daily.
  Other Names: No other names.
  Arms: Ferrofumerat (iron supplementation)

SUMMARY:
Hemoboost is a registered natural product containing specially processed haemolysed haemoglobin and iron dextran. It is marketed for human use on the basis of many years' use and documented effect in veterinary medicine. Iron dextran was introduced for use in human medicine in 1954.

Krauterblut is a registered natural product made from a number of herbs where the active substance is ferrous gluconate. Both drugs have been available for a number of years and have become increasingly popular among patients and healthcare staff due to a reduction in adverse effects.

The objective of this study is to determine the effect and adverse effects of the natural products Hemoboost and Kräuterblut compared with the usually administered ferrous sulphate in knee arthroplasty.

DETAILED DESCRIPTION:
Hip and knee arthroplasties are performed with increasing frequency in the western world, and in Denmark approximately 12,000 operations are performed annually (2/1000/year). The perioperative and postoperative blood loss generally constitutes ½ -1½ litres which is frequently associated with symptom-producing anaemia which obstructs mobilisation and increases the risk of complications.

Postoperative iron supplementation for a period of up to 12 weeks is therefore a frequently adopted practice. However, there is no consensus or evidence that support postoperative iron supplementation and the effects of iron deficiency are unclear. It is well-known that iron supplementation causes gastrointestinal adverse effects in up to 25% of cases.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* ASA group I-II

Exclusion Criteria:

* malignant disorder
* chronic renal insufficiency
* urinary tract infection
* haemorrhagic diathesis
* haemoglobin < 7 mmol/l
* dementia or mental disorder incompatible with survey participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2006-05; Primary Completion 2006-12 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Haemoglobin concentration | 3 months
  Determine whether peroral iron substitution of Hemo-Boost or Krauterblut results in the same increase of haemoglobin concentration as the usually administered ferrous sulphate.
  To study the adverse effects of the natural products Hemo-Boost and Krauterblut compared with ferrous sulphate in knee arthroplasty.

SECONDARY OUTCOMES:
Pain measurement | 3 months
  Pain scores on the Visual Analog Scale.
Consumption af analgesics | 3 months
Healing of ulcer | 3 months
Basic need for facilities | 3 months
Level of activity | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Sten Rasmussen, M.D.Sci., Principal Investigator — Orthopaedic Division, North Denmark Region, Aalborg University Hospital, Denmark; Søren Lundbye-Christensen, Ph.d., Study Chair — Aalborg University; Mogens B. Joergensen, M.D., Study Chair — Orthopaedic Division, North Denmark Region, Aalborg University Hospital, Denmark; Ole Simonsen, M.D., Study Chair — Orthopaedic Division, North Denmark Region, Aalborg University Hospital, Denmark
Locations (1):
- Frederikshavn Hospital, Aalborg Hospital/Aarhus University, Frederikshavn, Denmark